CLINICAL TRIAL: NCT00005933
Title: Cognitive Function in Leukocyte Disorders
Brief Title: Learning and Behavior Problems in Children With Chronic Granulomatous Disease and Related Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000164; 00-I-0164
Record Dates: First submitted 2000-07-04; First posted 2000-07-05 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-07

CONDITIONS: Chediak Higashi Syndrome; Chronic Granulomatous Disease; Job's Syndrome; Leukocyte Disorder
Keywords: Chronic Disease; Pediatric; Pulmonary; Intelligence; Coping; Chronic Illness; Learning
MeSH Terms: conditions — Chediak-Higashi Syndrome; Granulomatous Disease, Chronic; Job Syndrome; Leukocyte Disorders; Chronic Disease

SUMMARY:
This study will try to determine what causes learning, behavioral and emotional problems in children with chronic granulomatous disease (GCD) and other phagocyte disorders. (Phagocytes are a type of white blood cell.) Children with these disorders have frequent severe infections that require hospitalization, sometimes for long periods of time. Many of them also have problems with school, learning, behavior, anxiety and depression. This study will explore whether these latter problems are a direct result of the illness itself or are a consequence of frequent, long hospitalizations, or are due to other factors. Test findings in these children will be compared with those of children with cystic fibrosis-another disease that causes frequent infections requiring prolonged hospitalization.

Patients age 2 or older with GCD or other phagocytic disorders or cystic fibrosis may be eligible for this study. Participants (or a parent or guardian) will complete questionnaires including personal information such as age, gender and marital status, a family medical history, and information on their illness. Patients will be given various psychological and intelligence tests, and they and their parents or guardians will be interviewed by a child psychiatrist. The tests and interviews take a total of about 5 hours and are given in two or three separate sessions.

The tests may reveal problems such as learning disorders, attention-deficit hyperactivity disorder, anxiety, or depression. If any of these problems are identified, appropriate referrals will be made for specialized services, such as special school placement, tutoring, or counseling.

DETAILED DESCRIPTION:
Leukocyte disorders are predominantly genetic diseases in which phagocytes fail to function normally resulting in recurrent infections. Children with these disorders are subject to recurrent, severe, often life-threatening infections and are hospitalized more frequently than their peers. Frequent hospitalization and chronic illness can affect growth, development, socialization, and educational opportunities.

Specifically, chronic granulomatous disease (CGD) is an inherited disorder in which phagocytes fail to generate an oxidative burst. In 26 patients followed at the NIH tested for behavioral problems at the request of a parent or staff member, we have observed a 23% rate of mild mental retardation. However, it is not clear whether this is due to CGD per se or the recurrent infections and hospitalizations. We seek to determine the prevalence of cognitive disabilities in children with CGD and other leukocyte disorders. We seek to determine whether abnormal leukocyte functioning may be related to specific behavioral phenotypes or impaired cognitive functioning. We also seek to clarify whether impaired cognitive functioning is related to the effects of frequent and prolonged hospitalization or other variables such as severity of illness in this population.

ELIGIBILITY:
INCLUSION CRITERIA

Presence of a confirmed diagnosis of CGD or other phagocytic disorder.

Age 2 or older.

English spoken in the home.

EXCLUSION CRITERIA

Unconfirmed phagocytic disorder.

Under age 2.

First language is other than English.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 2000-06; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Batshaw ML. Mental retardation. Pediatr Clin North Am. 1993 Jun;40(3):507-21. doi: 10.1016/s0031-3955(16)38547-9. PMID 8493062
- [Background] Boyle IR, di Sant'Agnese PA, Sack S, Millican F, Kulczycki LL. Emotional adjustment of adolescents and young adults with cystic fibrosis. J Pediatr. 1976 Feb;88(2):318-26. doi: 10.1016/s0022-3476(76)81011-6. PMID 1249700
- [Background] Eliez S, Reiss AL. Genetics of childhood disorders: XI. Fragile X syndrome. J Am Acad Child Adolesc Psychiatry. 2000 Feb;39(2):264-6. doi: 10.1097/00004583-200002000-00029. No abstract available. PMID 10673840